CLINICAL TRIAL: NCT05056558
Title: Efficacy and Safety of Baricitinib in Patients With Moderate and Severe COVID-19 - A Multicenter Randomized Double Blind Placebo Controlled Clinical Trial in Bangladesh
Brief Title: Efficacy and Safety of Baricitinib in Patients With Moderate and Severe COVID-19
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Incepta Pharmaceuticals Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021/BR8/P3/01
Record Dates: First submitted 2021-09-20; First posted 2021-09-24 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — baricitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baricitinib (Experimental): Continued SOC together with oral 4 mg Baricitinib from day 1 to day 14
  Interventions: Drug: Baricitinib
- Placebo (Placebo Comparator): Continued SOC according as mentioned in operational definition in the protocol
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Baricitinib — Continued standard of care (SOC) together with oral 4 mg Baricitinib tablet from day 1 to day 14
  Other Names: Baricent
  Arms: Baricitinib
Drug: Placebo — Continued standard of care (SOC) together with oral placebo tablet from day 1 to day 14
  Other Names: Given Orally
  Arms: Placebo

SUMMARY:
This is multicenter clinical trial to evaluate efficacy and safety of Baricitinib in treatment for COVID-19. This trial will compare Baricitinib, a drug recommended for Rheumatoid Arthritis, against standard of care, to assess its relative effectiveness against COVID-19. By enrolling patients in multiple centers, this trial aims to recruit more patients to evaluate whether this drug slow disease progression or improve survival. Currently no effective therapeutics treatment or vaccine is available in the world for this highly transmissible respiratory borne infection, Covid-19. A number of drug trials are ongoing to measure the efficacy of the drug against the virus. Bangladesh as a resource limited country with limitation to provided health care services to the huge number of Covid-19 patients who will need hospitalization will be benefited from this study. There is no physical, psychological, social, legal risk in this study. The trial therapeutic will be approved form the Directorate of drug Administration (DGDA), Bangladesh.

ELIGIBILITY:
Inclusion Criteria:

* SARS-Co-V2 positivity to the nasal-swab by reverse-transcriptase-polymerase chain- reaction (RT-PCR) assay tested by the local diagnostic laboratory
* Age >18 years
* Presence of any symptoms suggestive of COVID-19, such as such as fever, fatigue, cough (with or without sputum production), shortness of breath, sore throat, nasal congestion, anorexia, malaise, or headache. Rarely, patients may also present with diarrhea, nausea, and vomiting
* Presence of radiological findings of pneumonia assessed by chest radiograph, computed tomography
* Moderate and severe COVID-19 as per previous definition national guideline/WHO
* Give informed written consent

Exclusion Criteria:

* Absolute lymphocyte count <500/mm3 and absolute neutrophil count of <1000/mm3 and Hemoglobin 8gm/dl or less
* Severe hepatic or renal impairment
* Live vaccine within 3 months prior to first dose of the drug
* Pregnancy
* Lactation
* Current malignancy or history of malignancies over the previous 5 years and/or history of malignancies in first degree relatives
* Transaminases values 5-fold higher than the upper normal limit
* Proven evidence of concomitant bacterial infections
* Clinical evidences suggestive of pulmonary tuberculosis, or past history and/or history of contact with TB patient
* Known hypersensitivity to Baricitinib
* Those who have received Tocilizumab previously

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Clinical status assessed by a 7-point ordinal scale on Day 14 | Day 1 to Day 14
  The ordinal scale is an assessment of the clinical status at a given study day. Each day, the worst(ie, lowest ordinal) score from the previous day will be recorded, ie, on Day 3, the lowest ordinal score from Day 2 is obtained and recorded for Day 2. The scale is as follows:
  1. Death
  2. Hospitalized, on invasive mechanical ventilation or ECMO
  3. Hospitalized, on non-invasive ventilation or high flow oxygen devices
  4. Hospitalized, requiring low flow supplemental oxygen
  5. Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise)
  6. Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care (other than per protocol Baricitinib administration)
  7. Not hospitalized

SECONDARY OUTCOMES:
The proportion of participants with treatment emergent adverse events | Day 1 to Day 28

OTHER OUTCOMES:
Time to clinical improvement (days): clinical improvement is defined as a ≥ 2-point improvement in clinical status (7-point ordinal scale) from Day 1 | Day 1 to Day 28
Time to ≥ 1-point improvement (days) from baseline clinical status | Day 1 to Day 28
Time to recovery: defined as an improvement in clinical status from a baseline score of 2 through 5 to a score of 6 or 7, or an improvement from a baseline score of 6 to a score of 7 | Day 1 to Day 28
Duration of oxygen therapy (days) | Day 1 to Day 28
Proportion of patients with shift in oxygen support status from baseline | Day 1 to Day 28
Duration of hospitalization (days) | Day 1 to Day 28
Number of patients with all-cause mortality at Day 28 | Day 1 to Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Md. Titu Miah, MBBS, FCPS, Principal Investigator — Dhaka Medical College; Md. Mujibur Rahman, MBBS, MD, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Dhaka Medical College, Mugda Medical College, Kuwait Bangladesh Friendship Government Hospital, Dhaka, Bangladesh